| Statistical Analysis Plan | |
|---|---|
| Title: Dietary Ketosis a Metabolic Sister to Calorie Restriction (CR): Fatty acids activate AMPK energy | |
| Title: Dietary Ketosis a Metabolic Sister to Calorie Restriction (CR): Fatty acids activate AMPK circuits modulating global methylation via the SAM/SAH axis | energy |
| Title: Dietary Ketosis a Metabolic Sister to Calorie Restriction (CR): Fatty acids activate AMPK circuits modulating global methylation via the SAM/SAH axis NCT03319173 | energy |
| circuits modulating global methylation via the SAM/SAH axis | <b>Cenergy</b> |
| circuits modulating global methylation via the SAM/SAH axis NCT03319173 | energy |

## Statistical Analyses Plan (SAP)

Aaron Rendahl, PhD

15 January, 2019

All analyses performed using R version 3.5.2 (2018-12-20). Standard citation is:

R Core Team (2018). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL <a href="https://www.R-project.org/">https://www.R-project.org/</a>.

## Analysis Plan

To assess differences between the control and experimental groups, a mixed model will be fit for each variable separately using both baseline (week 0) and post program (week 12) values for each subject. Models will include week, group, and their interaction as fixed effects, gender as a covariate, and subject as a random effect. To assess significant differences, we will use the difference at week 12 adjusted for the baseline difference, and will report p-values, least squares means, and 95% confidence intervals. Further analysis of treatment effects over time will be examined by comparing the within-group differences over time.

Variables that will be modeled are HgA1c, fasting insulin, fasting glucose, NMR particle size testing, SAM/SAH ratio test and whole blood histamine from the methylation profile, and the cognitive measures, the Ray Auditory Verbal Learning Task, BVMT-R, and MoCA. Additionally, blood ketones and fasting triglycerides.

NOTE: For blood ketones and fasting triglycerides, we planned to use all measured weeks (0, 3, 6, 9, and 12) but so far we are only using weeks 0 and 12.

Variables will be checked for normality using the Box-Cox method and by viewing applots on the residuals. Variables that are more normally distributed after a log transformation will be transformed and ratios will be reported instead of raw differences.

After checking the Box-Cox results, all should be log-transformed except MoCA and LP-IR and SAH.

For consistency, LP-IR is log-transformed too, it's not that much better on the original scale.



Figure 1: Boxplots for each variable, separated by timepoint and treatment group, with jittered points showing the individual data points. Variables that were log-transformed for analysis are plotted on the log-scale.

## Results

The first table shows the difference (as either a ratio or a raw difference) of week 12 compared to week 1, between the two groups, along with 95% confidence intervals and p-values. That is, for a ratio, it is (week 12 / week 1 for Treatment) / (week 12 / week 1 for Control).

The second table shows the estimated marginal means (also known as least square means) for each combination, as back-transformed from the model with a log transformation was used, along with 95% confidence intervals.

Finally, for evaluation of how this affects individuals, the mean and standard deviation, as well as the median, quantiles, and ranges for the differences (or ratios) are reported for each group.

These tables are also included as csv files (named diffs, estimates, and groups).

Table 1: Estimated differences in the change from day 0 to day 12 between treatment and control groups, as either an absolute difference or a ratio (if the variable was log-transformed). A negative change (or ratio less than 1 1) means the treatment group decreased relative to the control group. Also included are 95% confidence intervals and p-values. All values are estimated from the linear mixed models.

| var | measure | estimate | SE | df | lower.CL | upper.CL | t.ratio p.value |
|---|---|---|---|---|---|---|---|
| MoCA | diff | 8.241 | 0.229 | 96 | 7.786 | 8.696 | 35.947 < 0.0001 |
| Small<br>LDL | ratio | 0.348 | 0.021 | 96 | 0.308 | 0.393 | -17.242 < 0.0001 |
| LP-IR | ratio | 0.461 | 0.027 | 96 | 0.410 | 0.518 | -13.114 < 0.0001 |
| Trig | ratio | 0.514 | 0.024 | 96 | 0.468 | 0.564 | -14.062 < 0.0001 |
| HDL | ratio | 1.165 | 0.024 | 96 | 1.119 | 1.213 | 7.547 < 0.0001 |
| Tri/HDL | ratio | 0.441 | 0.024 | 96 | 0.395 | 0.491 | -14.967 < 0.0001 |
| Insulin | ratio | 0.444 | 0.022 | 96 | 0.402 | 0.491 | -16.039 < 0.0001 |
| Glucose | ratio | 0.747 | 0.015 | 96 | 0.719 | 0.777 | -14.776 < 0.0001 |
| HOMA-IR | ratio | 0.332 | 0.020 | 96 | 0.296 | 0.373 | -18.750 < 0.0001 |
| HgA1c | ratio | 0.867 | 0.007 | 96 | 0.853 | 0.881 | -17.742 < 0.0001 |
| Weight | ratio | 0.865 | 0.007 | 96 | 0.850 | 0.879 | -17.240 < 0.0001 |
| BFM | ratio | 0.752 | 0.022 | 96 | 0.709 | 0.798 | -9.578 < 0.0001 |
| VLDL | ratio | 0.514 | 0.024 | 96 | 0.468 | 0.564 | -14.062 < 0.0001 |
| SAM | ratio | 1.037 | 0.006 | 80 | 1.025 | 1.049 | 6.302 < 0.0001 |
| SAH | ratio | 0.925 | 0.008 | 80 | 0.909 | 0.942 | -8.730 < 0.0001 |
| SAM/SAH | ratio | 1.130 | 0.013 | 80 | 1.104 | 1.156 | 10.412 < 0.0001 |

| var | measure | estimate | SE | df | lower.CL | upper.CL | t.ratio p.value |
|---|---|---|---|---|---|---|---|
| Adenosine | ratio | 1.122 | 0.014 | 80 | 1.096 | 1.149 | 9.556 < 0.0001 |

Table 2: Estimated average values and 95% confidence intervals for each variable for day 0 and day 12 for both the treatment and control groups, as estimated by the linear mixed models, and back-transformed for variables that were first log transformed.

| var | time | Group | emmean | SE | df | lower.CL | upper.CL |
|---|---|---|---|---|---|---|---|
| MoCA | 1 | Control | 20.437 | 0.216 | 124.653 | 20.009 | 20.864 |
| MoCA | 2 | Control | 20.217 | 0.216 | 124.653 | 19.789 | 20.644 |
| MoCA | 1 | Treated | 20.358 | 0.221 | 124.653 | 19.921 | 20.794 |
| MoCA | 2 | Treated | 28.378 | 0.221 | 124.653 | 27.942 | 28.815 |
| Small LDL | 1 | Control | 522.881 | 54.254 | 103.438 | 425.634 | 642.346 |
| Small LDL | 2 | Control | 588.076 | 61.019 | 103.438 | 478.704 | 722.436 |
| Small LDL | 1 | Treated | 705.506 | 74.713 | 103.438 | 571.862 | 870.382 |
| Small LDL | 2 | Treated | 276.244 | 29.254 | 103.438 | 223.915 | 340.802 |
| LP-IR | 1 | Control | 48.608 | 2.575 | 128.164 | 43.771 | 53.979 |
| LP-IR | 2 | Control | 50.663 | 2.684 | 128.164 | 45.622 | 56.261 |
| LP-IR | 1 | Treated | 66.939 | 3.619 | 128.164 | 60.148 | 74.497 |
| LP-IR | 2 | Treated | 32.135 | 1.737 | 128.164 | 28.875 | 35.763 |

| var | time | Group | emmean | SE | df | lower.CL | upper.CL |
|---------|------|---------|---------|--------|---------|----------|----------|
| Trig | 1 | Control | 121.520 | 7.818 | 108.453 | 106.972 | 138.046 |
| Trig | 2 | Control | 131.728 | 8.474 | 108.453 | 115.958 | 149.643 |
| Trig | 1 | Treated | 156.660 | 10.286 | 108.453 | 137.543 | 178.434 |
| Trig | 2 | Treated | 87.229 | 5.727 | 108.453 | 76.585 | 99.353 |
| HDL | 1 | Control | 51.364 | 1.836 | 102.794 | 47.848 | 55.138 |
| HDL | 2 | Control | 48.900 | 1.748 | 102.794 | 45.553 | 52.493 |
| HDL | 1 | Treated | 46.953 | 1.713 | 102.794 | 43.675 | 50.476 |
| HDL | 2 | Treated | 52.097 | 1.901 | 102.794 | 48.461 | 56.007 |
| Tri/HDL | 1 | Control | 2.366 | 0.200 | 105.245 | 2.001 | 2.798 |
| Tri/HDL | 2 | Control | 2.694 | 0.228 | 105.245 | 2.278 | 3.186 |
| Tri/HDL | 1 | Treated | 3.337 | 0.288 | 105.245 | 2.812 | 3.959 |
| Tri/HDL | 2 | Treated | 1.674 | 0.145 | 105.245 | 1.411 | 1.987 |
| Insulin | 1 | Control | 10.595 | 0.733 | 108.241 | 9.237 | 12.152 |
| Insulin | 2 | Control | 11.252 | 0.778 | 108.241 | 9.810 | 12.905 |
| Insulin | 1 | Treated | 15.518 | 1.096 | 108.241 | 13.491 | 17.849 |
| Insulin | 2 | Treated | 7.323 | 0.517 | 108.241 | 6.367 | 8.424 |

| var | time | Group | emmean | SE | df | lower.CL | upper.CL |
|---------|------|---------|---------|-------|---------|----------|----------|
| Glucose | 1 | Control | 106.208 | 2.036 | 122.629 | 102.252 | 110.316 |
| Glucose | 2 | Control | 109.606 | 2.102 | 122.629 | 105.523 | 113.846 |
| Glucose | 1 | Treated | 111.368 | 2.179 | 122.629 | 107.136 | 115.767 |
| Glucose | 2 | Treated | 85.903 | 1.681 | 122.629 | 82.639 | 89.296 |
| HOMA-IR | 1 | Control | 2.778 | 0.222 | 108.485 | 2.372 | 3.254 |
| HOMA-IR | 2 | Control | 3.045 | 0.243 | 108.485 | 2.600 | 3.566 |
| HOMA-IR | 1 | Treated | 4.267 | 0.347 | 108.485 | 3.632 | 5.014 |
| HOMA-IR | 2 | Treated | 1.553 | 0.126 | 108.485 | 1.322 | 1.825 |
| HgA1c | 1 | Control | 5.730 | 0.046 | 121.498 | 5.640 | 5.821 |
| HgA1c | 2 | Control | 5.820 | 0.047 | 121.498 | 5.728 | 5.912 |
| HgA1c | 1 | Treated | 5.897 | 0.048 | 121.498 | 5.802 | 5.993 |
| HgA1c | 2 | Treated | 5.191 | 0.042 | 121.498 | 5.108 | 5.276 |
| Weight | 1 | Control | 209.187 | 5.712 | 97.248 | 198.151 | 220.836 |
| Weight | 2 | Control | 210.595 | 5.751 | 97.248 | 199.486 | 222.323 |
| Weight | 1 | Treated | 230.042 | 6.411 | 97.248 | 217.663 | 243.125 |
| Weight | 2 | Treated | 200.232 | 5.581 | 97.248 | 189.457 | 211.620 |

| var | time | Group | emmean | SE | df | lower.CL | upper.CL |
|------|------|---------|--------|-------|---------|----------|----------|
| BFM | 1 | Control | 79.578 | 3.470 | 106.408 | 72.988 | 86.763 |
| BFM | 2 | Control | 79.353 | 3.460 | 106.408 | 72.782 | 86.517 |
| BFM | 1 | Treated | 90.562 | 4.030 | 106.408 | 82.915 | 98.915 |
| BFM | 2 | Treated | 67.947 | 3.024 | 106.408 | 62.209 | 74.214 |
| VLDL | 1 | Control | 24.304 | 1.564 | 108.453 | 21.394 | 27.609 |
| VLDL | 2 | Control | 26.346 | 1.695 | 108.453 | 23.192 | 29.929 |
| VLDL | 1 | Treated | 31.332 | 2.057 | 108.453 | 27.509 | 35.687 |
| VLDL | 2 | Treated | 17.446 | 1.145 | 108.453 | 15.317 | 19.871 |
| SAM | 1 | Control | 89.365 | 2.646 | 79.783 | 84.252 | 94.789 |
| SAM | 2 | Control | 88.177 | 2.611 | 79.783 | 83.131 | 93.529 |
| SAM | 1 | Treated | 87.723 | 2.535 | 79.783 | 82.821 | 92.915 |
| SAM | 2 | Treated | 89.784 | 2.594 | 79.783 | 84.767 | 95.099 |
| SAH | 1 | Control | 19.448 | 0.319 | 85.209 | 18.825 | 20.093 |
| SAH | 2 | Control | 19.566 | 0.321 | 85.209 | 18.938 | 20.214 |
| SAH | 1 | Treated | 19.616 | 0.314 | 85.209 | 19.002 | 20.250 |
| SAH | 2 | Treated | 18.257 | 0.292 | 85.209 | 17.685 | 18.847 |

| var | time | Group | emmean | SE | df | lower.CL | upper.CL |
|-----------|------|---------|--------|-------|--------|----------|----------|
| SAM/SAH | 1 | Control | 4.595 | 0.200 | 80.482 | 4.214 | 5.010 |
| SAM/SAH | 2 | Control | 4.491 | 0.195 | 80.482 | 4.119 | 4.896 |
| SAM/SAH | 1 | Treated | 4.472 | 0.190 | 80.482 | 4.110 | 4.866 |
| SAM/SAH | 2 | Treated | 4.938 | 0.209 | 80.482 | 4.538 | 5.372 |
| Adenosine | 1 | Control | 22.524 | 0.482 | 85.700 | 21.587 | 23.503 |
| Adenosine | 2 | Control | 21.475 | 0.459 | 85.700 | 20.581 | 22.407 |
| Adenosine | 1 | Treated | 21.837 | 0.456 | 85.700 | 20.950 | 22.762 |
| Adenosine | 2 | Treated | 23.363 | 0.488 | 85.700 | 22.413 | 24.352 |

Table 3: Descriptive statistics on the changes for each variable from day 0 to day 12 for each group, including mean, standard deviation, median, quartiles, and ranges. Changes were first computed for each individual as an absolute difference, or a ratio for variables that were log-transformed.

| var | Group | measure | mean | sd | min | Q1 | median | Q3 | max |
|---|---|---|---|---|---|---|---|---|---|
| MoCA | Control | diff | -0.220 | 0.954 | -3.000 | -1.000 | 0.000 | 0.000 | 2.000 |
| MoCA | Treated | diff | 8.021 | 1.296 | 5.000 | 7.000 | 8.000 | 9.000 | 11.000 |
| Small<br>LDL | Control | ratio | 1.142 | 0.230 | 0.891 | 1.040 | 1.058 | 1.147 | 2.037 |
| Small<br>LDL | Treated | ratio | 0.422 | 0.164 | 0.134 | 0.318 | 0.398 | 0.524 | 1.000 |
| LP-IR | Control | ratio | 1.055 | 0.174 | 0.703 | 1.028 | 1.063 | 1.094 | 1.935 |

| var | Group | measure | mean | sd | min | Q1 | median | Q3 | max |
|---|---|---|---|---|---|---|---|---|---|
| LP-IR | Treated | ratio | 0.513 | 0.172 | 0.164 | 0.394 | 0.517 | 0.613 | 0.931 |
| Trig | Control | ratio | 1.105 | 0.257 | 0.767 | 1.031 | 1.048 | 1.108 | 2.306 |
| Trig | Treated | ratio | 0.577 | 0.145 | 0.291 | 0.501 | 0.579 | 0.683 | 0.893 |
| HDL | Control | ratio | 0.955 | 0.076 | 0.596 | 0.932 | 0.959 | 0.983 | 1.190 |
| HDL | Treated | ratio | 1.117 | 0.131 | 0.833 | 1.050 | 1.101 | 1.150 | 1.587 |
| Tri/HDL | Control | ratio | 1.169 | 0.317 | 0.787 | 1.039 | 1.100 | 1.178 | 2.416 |
| Tri/HDL | Treated | ratio | 0.526 | 0.157 | 0.232 | 0.415 | 0.520 | 0.626 | 0.986 |
| Insulin | Control | ratio | 1.068 | 0.116 | 0.806 | 1.016 | 1.061 | 1.128 | 1.342 |
| Insulin | Treated | ratio | 0.498 | 0.163 | 0.198 | 0.387 | 0.484 | 0.576 | 0.928 |
| Glucose | Control | ratio | 1.034 | 0.059 | 0.898 | 0.991 | 1.044 | 1.063 | 1.176 |
| Glucose | Treated | ratio | 0.777 | 0.088 | 0.438 | 0.735 | 0.788 | 0.839 | 0.913 |
| HOMA-IR | Control | ratio | 1.105 | 0.139 | 0.859 | 1.033 | 1.129 | 1.181 | 1.553 |
| HOMA-IR | Treated | ratio | 0.391 | 0.143 | 0.101 | 0.303 | 0.374 | 0.469 | 0.839 |
| HgA1c | Control | ratio | 1.016 | 0.037 | 0.943 | 0.983 | 1.017 | 1.036 | 1.131 |
| HgA1c | Treated | ratio | 0.881 | 0.037 | 0.742 | 0.869 | 0.882 | 0.899 | 0.947 |
| Weight | Control | ratio | 1.007 | 0.018 | 0.949 | 0.994 | 1.011 | 1.018 | 1.040 |

| var | Group | measure | mean | sd | min | Q1 | median | Q3 | max |
|---|---|---|---|---|---|---|---|---|---|
| Weight | Treated | ratio | 0.872 | 0.049 | 0.743 | 0.841 | 0.868 | 0.903 | 1.003 |
| BFM | Control | ratio | 1.000 | 0.068 | 0.548 | 0.996 | 1.009 | 1.024 | 1.065 |
| BFM | Treated | ratio | 0.762 | 0.124 | 0.378 | 0.711 | 0.780 | 0.843 | 1.010 |
| VLDL | Control | ratio | 1.105 | 0.257 | 0.767 | 1.031 | 1.048 | 1.108 | 2.306 |
| VLDL | Treated | ratio | 0.577 | 0.145 | 0.291 | 0.501 | 0.579 | 0.683 | 0.893 |
| SAM | Control | ratio | 0.987 | 0.031 | 0.876 | 0.975 | 0.987 | 1.000 | 1.054 |
| SAM | Treated | ratio | 1.024 | 0.020 | 0.977 | 1.011 | 1.025 | 1.035 | 1.068 |
| SAH | Control | ratio | 1.007 | 0.040 | 0.975 | 0.990 | 1.000 | 1.011 | 1.230 |
| SAH | Treated | ratio | 0.932 | 0.041 | 0.860 | 0.899 | 0.927 | 0.963 | 1.011 |
| SAM/SAH | Control | ratio | 0.979 | 0.051 | 0.780 | 0.966 | 0.982 | 1.006 | 1.057 |
| SAM/SAH | Treated | ratio | 1.105 | 0.058 | 1.004 | 1.068 | 1.099 | 1.137 | 1.296 |
| Adenosine | Control | ratio | 0.954 | 0.046 | 0.870 | 0.916 | 0.953 | 0.973 | 1.056 |
| Adenosine | Treated | ratio | 1.072 | 0.066 | 0.947 | 1.040 | 1.053 | 1.100 | 1.263 |